CLINICAL TRIAL: NCT00721890
Title: Phase II Study: Green Tea Intake for the Maintenance of Complete Remission in Women With Advanced Ovarian Carcinoma
Brief Title: Green Tea Intake for the Maintenance of Complete Remission in Women With Advanced Ovarian Carcinoma
Acronym: DBGT-OC-CR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Cancer Research Society (Other)
Responsible Party: Principal Investigator, Bernard Têtu, Professor, MD, CHU de Quebec-Universite Laval
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: SC-126639
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Ovarian Carcinoma
Keywords: chemoprevention; green tea; relapse free-survival; proteases
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Dietary Supplement: Double-Brewed Green Tea

INTERVENTIONS:
Dietary Supplement: Double-Brewed Green Tea — liquid, 4 celsius; 500 mL ID, 3 hours after meals and 1 hour before next meal; duration: to the first of the following events: 18 months or relapse
  Other Names: DBGT

SUMMARY:
Green tea is extracted from steam treated leaves, allowing the preservation of catechins, the active elements of the infusion. Catechins are recognized for their anti-cancer activity. Catechins act on the capacity of cancer to disseminate to other organs because of their anti-protease action. Proteases are proteins capable of digesting the cancer environment and facilitating the progression of cancer cells to blood vessels which will bring them to distant organs. We know that ovarian cancer responds well to the initial treatment of chemotherapy but tends to recur rapidly. We intend to provide green tea with higher concentrations of catechins to women with complete remission of their ovarian cancer in an attempt to delay cancer relapse. We also intend to identify, with molecular technologies, the proteases involved in ovarian cancer recurrence and response to catechins. Our objective is to test the hypothesis that green tea intake may delay ovarian cancer recurrence and to develop tools to predict which women will best benefit of the addition of green tea to their initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with ovarian serous carcinoma FIGO stage III or IV
* patients showing complete response after oncological surgery and chemotherapy (paclitaxel-carboplatin, minimum 5 cycles, maximum 8 cycles), complete response being defined as 1) a negative complete physical examination 2) Serum CA-125 levels inferior to 35 U/mL 3) no evidence of diseased assessed by abdomino-perineal CT-scan
* patients refraining from drinking tea other than provided by the study
* patients who may absorb liquids orally
* patients without any other malignancy (except for non-melanoma skin cancer)
* patients not involved in an other study
* patients who signed up informed consent form.

Exclusion Criteria:

* exclusion criteria are implicit from inclusion criteria.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
time to relapse | 36 months

SECONDARY OUTCOMES:
toxicity | 14th and 28th patients recruted and PRN

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Têtu, MD, Principal Investigator — Laval University; Isabelle Bairati, MD, Principal Investigator — Laval University; Marie Plante, MD, Study Chair — Laval University; Laurent Bazinet, PhD, Study Chair — Laval University; Dimcho Bachvarov, PhD, Study Chair — Laval University
Locations (1):
- Centre Hospitalier Universitaire de Québec, Hôtel-Dieu de Québec, Québec, Quebec, Canada

REFERENCES:
- [Derived] Trudel D, Labbe DP, Araya-Farias M, Doyen A, Bazinet L, Duchesne T, Plante M, Gregoire J, Renaud MC, Bachvarov D, Tetu B, Bairati I. A two-stage, single-arm, phase II study of EGCG-enriched green tea drink as a maintenance therapy in women with advanced stage ovarian cancer. Gynecol Oncol. 2013 Nov;131(2):357-61. doi: 10.1016/j.ygyno.2013.08.019. Epub 2013 Aug 27. PMID 23988418